CLINICAL TRIAL: NCT00945347
Title: Does a Nasal Instillation of Miglustat Normalize the Nasal Potential Difference in Cystic Fibrosis Patients Homozygous for the F508del Mutation? A Randomized, Double Blind Placebo-controlled Study.
Brief Title: Does a Nasal Instillation of Miglustat Normalize the Nasal Potential Difference in Cystic Fibrosis Patients ?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Patrick Lebecque, MD, PhD, Cliniques universitaires Saint Luc (Université Catholique de Louvain)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MIG-99
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; miglustat; nasal instillation; nasal potential difference
MeSH Terms: conditions — Cystic Fibrosis | interventions — miglustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Baseline (No Intervention): Visit 1
- Miglustat (Active Comparator): Nasal instillation of Miglustat (visit 2 or 3)
  Interventions: Drug: Miglustat
- Placebo (Placebo Comparator): Nasal instillation of placebo (visit 3 or 2)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Miglustat — Nasal instillation of miglustat
  Arms: Miglustat
Drug: Placebo — Nasal instillation of placebo matching in appearance with the Miglustat instillation
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate within a short delay the effect of nasal instillation of Miglustat on nasal potential difference in cystic fibrosis patients homozygous for the F508del mutation.

DETAILED DESCRIPTION:
Miglustat is an inhibitor of α-glucosidases and other enzymes. Oral miglustat is currently marketed in Europa and US for the treatment of Gaucher type 1 patients for whom enzyme replacement treatment is not an option.

Gastro-intestinal side effects are common with this formulation. This medication has been shown to have a beneficial effect both on Cl- an Na+ transports in cystic fibrosis epithelial cells. In addition, a single airway delivery of low-dose Miglustat normalizes nasal potential difference (NPD) in F508del cystic fibrosis mice. NPD abnormalities specific of CF patients are considered to reflect the primary defect of CFTR protein so that any curative treatment is expected to correct them at least partially.

In the field of respiratory pharmacology, it is a general rule that the inhaled route is to be favoured whenever possible : it is usually more effective despite much lower doses and systemic absorption (which also implies lower costs and improved tolerance).

The aim of this study is to investigate the effect of a single local administration of Miglustat on NPD measurements in CF patients homozygous for the F508del mutation.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis patients homozygous for the F508del mutation as confirmed by genetic test
* Aged 14 years and older
* Male or female (non-pregnant women who are to remain non-pregnant for 3 months after the end of the study)
* FEV1 > 50% of predicted normal

Exclusion Criteria:

* Acute respiratory tract infection or pulmonary exacerbation requiring antibiotic intervention within 2 weeks of visit 1
* Any condition prohibiting the correct measurement of the NPD such as respiratory tract infection
* Active or passive smoking
* Allergic chronic rhinitis
* History of significant lactose intolerance
* History of neuropathy
* History of cataracts or known increased risk of cataract formation
* Hypersensitivity to miglustat or any excipients
* Planned treatment or treatment with another investigational drug or therapy within 1 month prior to randomisation

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
change in response to Chloride-free solution and isoproterenol ( reflecting chloride transport) | change from baseline ( visit 1) and placebo to miglustat instillation

SECONDARY OUTCOMES:
change in basal voltage value and in amiloride response ( reflecting sodium transport) | change from baseline (visit1) and placebo to miglustat instillation

CONTACTS AND LOCATIONS:
Overall Officials: Patrick LEBECQUE, MD, PhD, Principal Investigator — Cliniques Universitaires St Luc (Université Catholique de Louvain ); Teresinha LEAL, MD, PhD, Principal Investigator — Cliniques Universitaires St. Luc ( Université Catholique de Louvain)
Locations (1):
- Cliniques Universitaires St Luc (Université Catholique de Louvain) 10 avenue Hippocrate, Brussels, Belgium

REFERENCES:
- [Background] Lubamba B, Lebacq J, Lebecque P, Vanbever R, Leonard A, Wallemacq P, Leal T. Airway delivery of low-dose miglustat normalizes nasal potential difference in F508del cystic fibrosis mice. Am J Respir Crit Care Med. 2009 Jun 1;179(11):1022-8. doi: 10.1164/rccm.200901-0049OC. Epub 2009 Mar 19. PMID 19299496
- [Background] Norez C, Noel S, Wilke M, Bijvelds M, Jorna H, Melin P, DeJonge H, Becq F. Rescue of functional delF508-CFTR channels in cystic fibrosis epithelial cells by the alpha-glucosidase inhibitor miglustat. FEBS Lett. 2006 Apr 3;580(8):2081-6. doi: 10.1016/j.febslet.2006.03.010. Epub 2006 Mar 10. PMID 16546175
- [Background] Noel S, Wilke M, Bot AG, De Jonge HR, Becq F. Parallel improvement of sodium and chloride transport defects by miglustat (n-butyldeoxynojyrimicin) in cystic fibrosis epithelial cells. J Pharmacol Exp Ther. 2008 Jun;325(3):1016-23. doi: 10.1124/jpet.107.135582. Epub 2008 Feb 28. PMID 18309088
- [Background] Norez C, Antigny F, Noel S, Vandebrouck C, Becq F. A cystic fibrosis respiratory epithelial cell chronically treated by miglustat acquires a non-cystic fibrosis-like phenotype. Am J Respir Cell Mol Biol. 2009 Aug;41(2):217-25. doi: 10.1165/rcmb.2008-0285OC. Epub 2009 Jan 8. PMID 19131642
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662